CLINICAL TRIAL: NCT01079767
Title: Advanced Hepatocellular Carcinoma on Child B Cirrhosis: Tolerance and Efficacy of Torisel® (Temsirolimus)
Brief Title: Temsirolimus in Treating Patients With Advanced Liver Cancer and Cirrhosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study treminated early according to DSMB recommendantions
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000666229; FFCD-0903; EUDRACT-2009-014443-36; EU-21004
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temsirolimus (Other): Temsirolimus
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: temsirolimus

SUMMARY:
RATIONALE: Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well temsirolimus works in treating patients with advanced liver cancer and cirrhosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the 3-month disease-control rate according to RECIST criteria in patients with advanced hepatocellular carcinoma and Child-Pugh class B cirrhosis.

Secondary

* To determine the 3-month objective response rate according to RECIST criteria in these patients.
* To determine the 1-month metabolic response rate on PET/CT scan in these patients.
* To determine the 1-month perfusion response rate on hepatic perfusion CT scan in these patients.
* To determine the time to progression in patients treated with this drug.
* To determine the progression-free survival of patients treated with this drug.
* To determine the overall survival of patients treated with this drug.
* To assess quality of life according to QLQ-C30 and QLQ-HCC18 questionnaires.
* To determine the clinical and biological tolerance of this drug in these patients.
* To determine the rate of m-TOR pathway activation and VEGF level.
* To evaluate the pharmacokinetics of this drug in select patients.

OUTLINE: This is a multicenter study.

Patients receive temsirolimus IV over 30-60 minutes on day 1. Treatment repeats once a week in the absence of disease progression or unacceptable toxicity. Patients also undergo fludeoxyglucose F 18 (FDG) positron emission tomography/computed tomography (PET/CT) scan and perfusion CT scan of the liver at baseline and periodically during study treatment.

Patients complete quality of life questionnaires (QLC-C30 and QLQ-HCC18) periodically. Some patients undergo blood and tissue sample collection periodically for pharmacological and laboratory studies.

After completion of study therapy, patients are followed for up to 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma (HCC) according to the European Association for the Study of the Liver (EASL) criteria

  * Advanced disease
  * Must be morphologically evaluable
* HCC not accessible to other treatment (e.g., surgery, radiofrequency, or chemoembolization) and can not benefit from antiangiogenic therapy
* CLIP score ≤ 3 (except for patients with tumors invading more than 50% of tumor volume)
* Child-Pugh cirrhosis score between B7 and B9, meeting the following criteria:

  * Diagnosed clinically, biologically (e.g., prothrombin time, platelets, or albumin), endoscopically (signs of portal hypertension) and morphologically (dysmorphic liver on ultrasound or CT scan), or by liver biopsy
* Not a candidate for transplantation and has not received a liver transplant

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Platelet count ≥ 50,000/mm^3
* Neutrophil count ≥ 1,500/mm^3
* Creatinine clearance ≥ 60 mL/min
* GFR ≥ 30 mL/min
* Serum cholesterol ≤ 350 mg/dL
* Triglycerides ≤ 300 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for more than 2 months after completion of study therapy
* No history of other cancer on treatment
* No cardiopulmonary disease impairment, including a history of stable or unstable angina or myocardial infarction
* No active infection except for viral hepatitis
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior inhibitors or inducers of P-glycoprotein, CYP3A4, or CYP3A5
* At least 4 weeks since prior surgery, radiotherapy (except radiotherapy to the bone), transarterial chemoembolization, immunotherapy, or other investigational drug for HCC
* At least 6 months since prior chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
3-month disease-control rate according to RECIST criteria | 2010

SECONDARY OUTCOMES:
3-month objective response rate according to RECIST criteria | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Decaens, MD, Principal Investigator — Centre Hospitalier Universitaire Henri Mondor; Christophe Duvoux, Principal Investigator — Centre Hospitalier Universitaire Henri Mondor
Locations (1):
- Centre Hospitalier Universitaire Henri Mondor, Créteil, France